CLINICAL TRIAL: NCT06653712
Title: Healthy Control Population für PAIS-ME/CFS: Studie Zur Evaluation möglicher Biomarker Und Untersuchungsmethoden für Die PAIS-ME/CFS-Diagnostik Bei Gesunden Probanden
Brief Title: Healthy Control Population for PAIS-ME/CFS: Study to Evaluate Possible Biomarkers and Methods for Examination of PAIS-ME/CFS Diagnostics in Healthy Volunteers
Acronym: HelP
Status: Not yet recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Charite University, Berlin, Germany (Other); Max-Planck Institut (Unknown); University Hospital Erlangen (Other)
Responsible Party: Sponsor
Other Study IDs: HelP
Record Dates: First submitted 2024-10-04; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Healthy Controls
Keywords: ME/CFS; Post-Covid; Biomarker
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy controls: Healthy participants between 10 and 25 years of age. We plan to recruit 5 to 10 participants per age group.
  Interventions: Diagnostic Test: Diagnostic Test

INTERVENTIONS:
Diagnostic Test: Diagnostic Test — The following clinical data sources are used:
  * Personal interview (anamnesis)
  * Physical examination
  * Questionnaires
  * Functional assessment
  * Imaging techniques
  The following biological materials are used:
  • Max. 30 ml of blood

SUMMARY:
Using the data from the HelP study, the underlying processes of the diseases ME/CFS and PAIS are to be researched and elucidated. The comparison of affected patients with healthy controls is intended to identify disease-specific patterns that could be related to the development or progression of the disease. The aim is to find a suitable biomarker for diagnostics and to develop therapeutic approaches.

DETAILED DESCRIPTION:
The underlying pathomechanisms of the diseases PAIS and ME/CFS are to be investigated and elucidated in more detail. The aim is to establish a cohort of healthy controls at our MRI Chronic Fatigue Center (MCFC). Within this cohort, the measurement instruments used so far in ME/CFS diagnostics will be validated. In addition, data material from this pool should be used for the statistical evaluations of various case-control studies of our center and our cooperation partners in order to find and develop a suitable biomarker for diagnostics and therapeutic approaches for PAIS and ME/CFS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy control subjects without a known medical diagnosis, except: asthma, allergies, neurodermatitis, if this does not require regular medication (self-disclosure)
* Age: 10 - 25 years
* Written declaration of consent or, in the case of minors, written declaration of consent from the participants and their legal representatives

Exclusion Criteria:

* Acute illnesses (e.g. infections) or major injuries
* Known chronic diseases (including psychological diagnoses) other than those mentioned above
* Surgery or blood transfusion in the last 3 months
* No intake of on-demand medication (e.g. painkillers) in the last 7 days before the date of the examination
* Pregnancy; Breastfeeding
* Limited legal capacity

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy controls are recruited via public relations
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Personal data | Measurement is taken at a single time point right after enrollment
  Name, date of birth, contact details
Clinical data | Measurement is taken at a single time point right after enrollment
  Sex, vaccination status, level of education, occupation, smoking and alcohol behavior, other addictive behavior, competitive sports
Physical assessment | Measurement is taken at a single time point right after enrollment
  weight and height will be combined to report BMI in kg/m^2
Heart rate | Measurement is taken at a single time point right after enrollment
  beats per minute
Blood pressure | Measurement is taken at a single time point right after enrollment
  in mmHg
Questionnaire data | Measurement is taken at a single time point right after enrollment
  Following questionnaires are rated on a scale: MBSQ, Chalder Fatigue Scale, PedsQL Fatigue, Bell Score, DSQ-PEM, SF-36, PedsQL, EQ5D, PHQ4, Compass31
YSR questionnaire | Measurement is taken at a single time point right after enrollment
  Open questions and questions to be rated on a scale
Imaging | Measurement is taken at a single time point right after enrollment
  OCT-A: Imaging of ocular fundus
Full blood count | Measurement is taken at a single time point right after enrollment
  CRP, Ferritin, Creatinin, GPT and Immunglobuline
Deformability Cytometer | Measurement is taken at a single time point right after enrollment
  Cell-deformation
Virology | Measurement is taken at a single time point right after enrollment
  EBV, CMV, HSV1, HSV2 and Sars CoV2 antibodies
Immunology | Measurement is taken at a single time point right after enrollment
  ANA, Cystatin C, dsDNA Ak
Endocrinology | Measurement is taken at a single time point right after enrollment
  TPO antibodies
B-cell phenotyping | Measurement is taken at a single time point right after enrollment
  Analysis of surface antigens using cytometry by time of flights (CyTOF)
Pain threshold | Measurement is taken at a single time point right after enrollment
  Measuring pressure tolerancy in Newton by means of an algometer at the iliotibial tract, phalanx distalis III, trapezius muscle in triplicates
Orthostasic Tolerance | Measurement is taken at a single time point right after enrollment
  blood pressure and heart rate are measured during the 10-minute standing test to determine orthostasic tolerance
Grip strength | Measurement is taken at a single time point right after enrollment
  Hand dynamometer test to assess grip strength in Newton
Smell test | Measurement is taken at a single time point right after enrollment
  Recognition of different substances